CLINICAL TRIAL: NCT01750671
Title: Influence Of Nutritional Status Of Patients In The Intensive Care Output On Long Term Fate
Acronym: FEEDING
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry); Baxter S.A.S (Unknown); University Hospital, Strasbourg, France (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0127
Record Dates: First submitted 2012-11-16; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Nutritional Status at the Release of ICU.
Keywords: ICU; Body composition; Nutrition; Survival; Morbidity

STUDY DESIGN:
Observational Model: Cohort

SUMMARY:
It is established that the surviving patients after a stay in the ICU are characterized by frequent malnutrition and morbidity and mortality. The main goal of this work is to study the relationship between nutritional statuses during ICU hospitalization, whatever its determinants, and quality of life, morbidity and mortality at one year.

The hypothesis of the study is that the presence of under nutrition is responsible for a 10% increase in crude mortality at one year (which would be respectively 30% for malnourished patients and 20% for non-malnourished patients).

DETAILED DESCRIPTION:
This is a multicenter cohort study of a 30-month follow-up on patients after a stay in ICU.

Nutritional parameters and evaluation of the quality of life will be collected during hospitalization and output during a visit to the Clinical Research Associate at 6 months and one year. Survival will be also noted. These parameters will be studied in comparative patients malnourished and non-malnourished.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, age greater than or equal to 18 years

  * Hospitalized more than 72 hours in the ICU
  * Requiring at least one support organ failure:

    1. Ventilatory support (invasive or noninvasive)
    2. Administration of catecholamines
    3. Extrarenal purification whatever technique
  * Affiliated to a social security system
  * Having given free, informed written consent

Exclusion Criteria:

* Patients with end-stage disease or for which a limitation of care was decided

  * Pregnant women
  * Patients with minor or under guardianship
  * Incapacitated adults and psychiatric inpatients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients malnourished and non-malnourished
Sampling Method: Probability Sample
Enrollment: 680 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | at one year

SECONDARY OUTCOMES:
Anxiety and depression | at inclusion, M6 and M12
Post-traumatic stress | at inclusion, M6 and M12
Quality of life | at M6 and M12
Degree of activity (Karnofsky questionnaire) | At M6 and M12
Weight | at inclusion, M6 and M12
Body mass index | at inclusion, M6 and M12
Albumin | at inclusion, M6 and M12
Orosomucoid | at inclusion, M6 and M12
Transthyretin (prealbumin) | at inclusion, M6 and M12
Body composition | at inclusion, M6 and M12

CONTACTS AND LOCATIONS:
Overall Officials: Noël CANO, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- Chu de Clermont-Ferrand, Clermont-Ferrand, France